CLINICAL TRIAL: NCT07392762
Title: Virtual Reality-Supported Exercise for Chronic Musculoskeletal Shoulder Disorders: a Feasibility Study (The V-RECS Study)
Brief Title: Virtual Reality-Supported Exercise for Chronic Musculoskeletal Shoulder Disorders: a Feasibility Study
Acronym: V-RECS
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Royal National Orthopaedic Hospital NHS Trust (Other)
Collaborators: SyncVR Medical (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 359174
Record Dates: First submitted 2026-01-15; First posted 2026-02-06 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2025-10

CONDITIONS: Shoulder Pain; Chronic Shoulder Pain; Musculoskeletal Shoulder Pain
Keywords: Virtual Reality; VR; Musculoskeletal Rehabilitation; Musculoskeletal Shoulder Pain; Chronic Shoulder Pain; Shoulder pain disorders
MeSH Terms: conditions — Shoulder Pain

STUDY DESIGN:
Intervention Model Description: The SyncVR FIT platform is designed to support unilateral or bilateral upper limb movement through a series of interactive games, tasks, and challenges delivered via a VR headset (PICO 4). Participants will use handheld controllers to engage with these activities, enabling the system to track upper limb motion.
  While wearing the headset, participants will see a virtual representation of their upper limbs-specifically their hands-within the VR environment. These virtual hands mirror the participants' real-time movements, enhancing the enhancing the sense of immersion and embodiment. A tablet device will be used by the intervention provider to monitor the session.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Virtual Reality Exercise Programme (Experimental): Consenting participants will attend three VR exercise sessions delivered by an upper limb physiotherapist at the Royal National Orthopaedic Hospital (RNOH), using the SyncVR FIT platform.
  The SyncVR FIT platform is designed to support unilateral or bilateral upper limb movement through a series of interactive games, tasks, and challenges delivered via a VR headset. Participants will use handheld controllers to engage with these activities, enabling the system to track upper limb motion. While wearing the headset, participants will see a virtual representation of their upper limbs-specifically their hands-within the VR environment. These virtual hands mirror the participants' real-time movements, enhancing the sense of immersion and embodiment. A tablet device will be used by the intervention provider to monitor the session.
  Interventions: Device: Virtual Reality

INTERVENTIONS:
Device: Virtual Reality — Participants will engage with a 30 minute shoulder exercise programme using the SyncVR platform. There will be three intervention sessions in total and they will be spaced out once per week for a period of three weeks.

SUMMARY:
People with long-term (chronic) shoulder disorders caused by injuries, overuse or conditions (such as arthritis) often need physiotherapy. This usually includes exercise therapy to help reduce pain, rebuild strength and make every day activities easier. However, it can be hard to stick to an exercise programme. People may stop due to pain, fear of making the symptoms worse or simply loosing motivation.

Virtual Reality (VR) is a technology that may help people say engaged with their exercise programmes by making exercises more enjoyable and interactive. When using a headset (similar to goggles), people can see and interact with a 3D virtual world. Their movement, especially their hands and arms, are shown as an 'avatar' (a virtual character) in this virtual world. Exercise can feel more like playing a game or engaging with tasks/challenges, rather than performing repetitive movements. This shift might help reduce focus on pain and increase motivation. VR also provides real-time feedback, helping people track their progress and adjust their movements instantly. This might lead to more accurate and consistent exercise performance and better recovery outcomes.

Before we can test whether VR exercise programmes are effective for people with chronic shoulder disorders, we firstly need to understand whether it is practical and acceptable for patients to use. This 'feasibility' study will therefore involve 20 patients with chronic shoulder disorders referred for physiotherapy at the Royal National Orthopaedic Hospital (RNOH) in Stanmore, United Kingdom. Participants will take part in three VR exercise sessions at the RNOH over a three-week period. Levels of pain, quality of life and sleep quality etc. will be measured before and after three weeks. Interviews will also be held up to two weeks after the final session to explore people's experiences and thoughts towards the VR exercise programme. The results will help us decide if a larger study should go ahead.

DETAILED DESCRIPTION:
Chronic shoulder disorders are long-lasting problems that cause pain, stiffness, or weakness in the shoulder. 'Chronic' means the condition has lasted for more than three months. These issues can make everyday tasks like reaching, lifting, or getting dressed, painful and difficult. Chronic shoulder disorders are very common. They affect people of all ages, but are more likely to occur in adults over 40. It is estimated that shoulder pain is one of the most frequent reasons people see a doctor for muscle or joint issues and up to 1 in 4 people may experience shoulder pain at some point in their lives.

There are several reasons someone might develop a chronic shoulder disorder. These include: repeated use or overuse of the shoulder (common in certain jobs or sports), injuries, such as a fall or sudden strain, wear and tear with age, poor posture and conditions like arthritis, frozen shoulder, or tendon problems (e.g., rotator cuff injuries).

Physiotherapy involving exercise is a key component for treating many chronic shoulder disorders. National guidelines recommend it as a fist line option before trying injections or surgery. These exercise programmes usually involve stretching, strengthening, range of movement exercises. There is also evidence that regular guided shoulder exercises are just as effective as surgery for some people. Studies show that people with large rotator cuff tears for example improve in pain, movement and quality of life over two years with results similar to those seen after surgery. However, even though exercise therapy can help many people with chronic shoulder disorders, several factors impact their effect and how well they work. These include staying consistent, using proper technique and sticking to a routine. People often struggle to follow shoulder exercise programmes, especially on their own, because of pain, low motivation or lack of feedback. Finding ways to overcome these barriers is important.

Immersive Virtual Reality (VR) is a technology that lets people experience and interact with a 3D virtual world using a headset. This virtual world can be designed for different settings and tasks, using sights and sounds to make it feel real. When wearing the headset, users can interact with the virtual world, where their movements (especially their hands and arms) are displayed on a screen as a virtual character (avatar), which they can use to control and navigate the environment to interact with the tasks/games. These capabilities mean that VR may offer benefits for rehabilitation. It can help increase motivation, give instant feedback, distract from pain, improve joint movement, and slowly expose people to difficult situations. One major barrier to recovery amongst people with chronic shoulder disorders is kinesiophobia, or the fear of movement. People often avoid certain helpful movements because they anticipate pain or injury, which leads to more stiffness, weakness, and pain. VR might help overcome this by combining both mental and physical strategies. For example, it can safely expose people to movements and distract them from pain. Another benefit of VR is that it turns exercise into more of a game. This can make it more fun, less repetitive, and more motivating. VR also gives real-time feedback on how someone is doing, helping them set goals and track their progress.

In recent years, VR has become more established for treating people with pain or nerve problems, such as stroke, burns, phantom limb pain, or Complex Regional Pain Syndrome (CRPS). Research into treating chronic muscle and joint (MSK) conditions, like chronic shoulder disorders, has not progressed as much as research for nerve-related conditions. However, Virtual Reality (VR) is now approved in the United States (US) for treating lower back pain, and recent studies show it might help improve outcomes for a variety of MSK problems. For people with shoulder issues, VR could help improve treatment by changing how exercises are delivered.

Although VR shows promise for helping people with chronic shoulder problems, there have only been a few small-scale studies so far. To build stronger evidence, there is first need to run small a smaller 'feasibility' study. This type of study helps to understand whether the treatment and the research methods are practical and acceptable for patients. This step is important before moving on to larger, more conclusive clinical trials in the future.

This is a feasibility study to evaluate the practicality of a VR-supported exercise programme delivered using the 'SyncVR FIT' platform (www.syncvrmedical.com) for patients with chronic MSK shoulder disorders within the context of an NHS outpatient setting. A process evaluation will be embedded to explore 'how' the intervention was implemented. The findings will be used to support the development of a future intervention/trial.

The secondary objectives will be to:

1. Evaluate the feasibility of recruitment, identifying the number of eligible patients, reasons for non-participation and consent rate
2. Evaluate intervention/protocol fidelity, including dropout rate, dose, adaptations and reach (who did and did not take part).
3. Identify the type and number of adverse events occurring during the intervention
4. Identify the completion rate of study outcome measures
5. Qualitatively explore acceptability, barriers, facilitators and perceptions towards implementation of the intervention from the perspectives of patients.

The study will take place over a 12-month period. Formal power calculations are not required as this is a feasibility study, hence 20 adult participants with chronic shoulder disorders will be recruited from a single centre at the Royal National Orthopaedics Hospital (RNOH) NHS Trust.

Inclusion criteria:

* Adult patients >18 years with diagnosed unilateral/ bilateral shoulder pain with/ without co-existing symptoms of instability and or stiffness (persisting > three months) generated from a Musculoskeletal origin
* Patients who have been referred for conservative management
* New or follow-up patients
* Patients presenting with MSK shoulder pain generated from traumatic and/or non-traumatic origins.
* Patients who provide informed, written consent to enter the study

Exclusion criteria

* Unable to provide informed consent
* On a waiting list for surgery and/or injections
* Referred for post-operative physiotherapy
* Shoulder pain not originating from an MSK aetiology (such as hemiplegia or peripheral nerve injury)
* Active history of seizures
* Other medical conditions deemed inappropriate for patients to participate e.g. visual impairment, unstable psychiatric illnesses.
* Shoulder pain associated with bone metastasis
* Currently taking part in any other upper limb research study
* Patients who do not adequately understand verbal explanations or written information given in English (or are not accompanied by an interpreter/family member).
* Patients who do not provide informed, written consent to enter the study

Screening, recruitment and consent:

Potential participants will be identified by the clinical care team and recruited from the RNOH therapies outpatients department, Stanmore.

Initial pre-screening of medical records will be conducted by the clinical care team, by reviewing patient lists on the hospital electronic notes system (EPIC).

Potential participants will be identified either in person during their outpatient appointments, or via telephone.

In person: Clinicians within the RNOH Therapies outpatient department will inform potential participants about the study during clinical appointments.

Via telephone: A member of the clinical care team will contact potentially eligible participants by phone to explain the study aims and objectives.

If interested, they will be given a Patient Information Sheet (PIS) to take home, posted or emailed depending on patient preference. The PIS provides contact details of the research team should they want to discuss the study further, either in person or via telephone when convenient to them. Alternatively, they can request a call from the research team, where verbal consent to initiate contact will be documented in the medical notes.

Study flyers will also be placed within the patient waiting/communal areas at the RNOH. The flyer will have contact details and a QR code, which can be scanned with a smartphone camera and will provide a link to the PIS and contact details of the research team.

Upon contact, a member of the research team will 1) determine interest, 2) provide a detailed overview of the study and 3) confirm eligibility and 4) provide an opportunity for questions.

Informed consent will be obtained once a full explanation of the study have been discussed. Consent will be obtained from a member of the research team as recorded on the sponsors delegation of responsibilities log either via telephone or in person.

Baseline visit (within 14 days of treatment visit 1):

The baseline visit will be combined with the screening visit whenever possible and subject to receiving informed consent and willingness and availability of participants. The following information will be collected:

1. Participant demographics (age, gender, ethnicity, employment status, social history, level of education)
2. Presenting complaint/Past medical history
3. History of motion sickness
4. Pain medication usage over past week
5. Shoulder range of movement
6. Subjective Shoulder pain intensity
7. Quality of life questionnaire
8. Shoulder pain and disability questionnaire
9. Sleep quality questionnaire

Intervention (treatment visit 1, 2 and 3):

Participants will be invited to take part in three VR exercise sessions, which will take place once per week for a period of three weeks. All sessions will take place within the therapies outpatient department at the RNOH and each session will last approximately one hour, although the actual time spent engaging with the exercise programme will be 30 minutes per session.

Each VR exercise session will broadly follow a similar format: 1) an explanation of the session activities/what to expect, 2) support to position the VR headset/prepare and 3) engage with a series of exercises delivered via the VR platform.

Upon wearing the VR headset, participants will see a virtual representation of their upper limbs, specifically their hands, within the virtual environment. These virtual hands mirror the participants' real-time movements, enhancing the sense of immersion and embodiment. A tablet device will be used by the intervention provider (physiotherapist) to monitor the session. A variety of engaging VR gaming tasks will be used to support upper limb rehabilitation by promoting range of movement (ROM), strength, motor control, and proprioception, such as boxing, archery and fruit picking. The session will be tailored to the goals/abilities of the participant and the tasks will intuitively progress though increasing levels of challenge/difficulty.

Subjective levels of pain intensity will be measured before and after each VR session and any adverse events occurring during the session will be recorded, as well as symptoms of cybersickness, which will be assessed using the Cybersickness in VR Questionnaire (CSQ-VR).

Follow-up Visit 1:

Follow-up one will take place via telephone or in person within 48 hours of treatment visit 3, regardless of whether participants completed all three sessions or not. The following information will be collected:

1. Pain medication usage over last week
2. Subjective shoulder pain intensity (NPRS)
3. Shoulder range of movement
4. Shoulder pain and disability questionnaire (SPADI)
5. Quality of life Questionnaire (EQ-5D-5L)
6. Quality of sleep questionnaire (PSQI)
7. Satisfaction questionnaire (QUEST)
8. Usability questionnaire (SUS)
9. Cybersickness in VR Questionnaire (CSQ-VR).

Follow-up two (optional):

Follow-up visit two will involve up to ten qualitative interviews with study participants in order to explore their experiences and perceptions towards implementation of the intervention. This visit will take place within two weeks after treatment visit 3. Qualitative interviews will be semi structured with the flexibility to explore concepts relating to the research question. Interviews will be conducted in-person, over the phone or by using MS Teams. Interviews will be audio recorded and transcribed word for word. Any personal identifiers (such as names or places) will be removed or changed from the transcripts prior to analysis.

Study endpoint:

Defined as the last patient visit.

Data analysis:

Quantitative data: No inferential statistics will be used as this is a feasibility study and no hypotheses are being tested, hence data will be analysed descriptively. The primary analysis will be to determine how feasible it is to recruit participants to the study and determine the dropout rate (defined as the proportion of people of who remained in in the study until the end), both of which will be described using frequencies and percentages. All other questionnaire data will also be summarised using averages where appropriate, or percentages depending on the type of data (continuous or categorical).

Qualitative data: Thematic analysis will identify and characterise empirical regularities in the data. Data will use Normalisation Process Theory (REF) to explain the acceptability (whether patients are willing to implement VR in clinical care) and the implementability (determinants / barriers / facilitators that shape whether VR can be implemented in practice). Factors that shape acceptability and implementability will be characterised in full.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients >18 years with diagnosed unilateral/ bilateral shoulder pain with/ without co-existing symptoms of instability and or stiffness (persisting > three months) generated from a Musculoskeletal origin
* Patients who have been referred for conservative management
* New or follow-up patients
* Sufficient English to understand written materials/verbal instruction/or accompanied by family/friends able to translate
* Patients who provide informed, written consent to enter the study

Exclusion Criteria:

* Unable to provide informed consent
* On a waiting list for surgery and/or injections
* Referred for post-operative physiotherapy
* Shoulder pain not originating from an MSK aetiology (such as hemiplegia or peripheral nerve injury)
* Active history of seizures
* Other relevant medical conditions deemed inappropriate for patients to participate e.g. visual impairment, unstable psychiatric illnesses.
* Shoulder pain associated with bone metastasis
* Currently taking part in any other upper limb research study
* Patients who do not adequately understand verbal explanations or written information given in English (or are not accompanied by an interpreter/family member).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2026-01-16 (Estimated); Primary Completion 2026-10-31 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Consent rate | During enrolment period
  The consent rate will be used as a measure of recruitment and will be defined as the number of participants who provide informed consent divided by the total number of patients screened for eligibility, ie: number of people who consented/number of people approached) x 100.
Dropout rate | From first treatment visit though completion of treatment (average of 3 weeks)
  The dropout rate will be defined as the percentage of participants who started the study, but did not complete all three treatment visits.

SECONDARY OUTCOMES:
Pain Intensity - Numeric Pain Rating Scale (NPRS) | * Baseline (Pre-intervention), * Immediately before and after each treatment session (up to 3 visits), * One follow-up 1 visit (within 48 hours of the last treatment session, average of 3 weeks)
  The NPRS is a validated, 11-item unidimensional numerical rating scale, with 0 representing 'no pain' and 10 representing 'worst imaginable pain' in the past 24 hours.
Shoulder Range of Movement | Baseline (pre-intervention) and at follow-up 1(within in 48 hours of final treatment session, average of 3 weeks).
  Shoulder ROM will be measured using a validated self-assessment questionnaire published by Yang et al 2015.
Disability - Shoulder Pain and Disability Index (SPADI) | Baseline (pre-intervention) and at follow-up 1(within in 48 hours of final treatment session, average of 3 weeks).
  The SPADI is a validated, self-administered questionnaire involving two dimensions (pain and functional activities) and 13 items. Scores can range between 0-100, where higher scores indicate worsening disability.
Quality of Life - EuroQol- 5 Dimension (EQ-5D-3L) | Baseline (pre-intervention) and at follow-up 1(within in 48 hours of final treatment session, average of 3 weeks).
  The EQ-5D-5L is a widely used, validated measure of health-related quality of life in terms of 5 dimensions (mobility, ability to self-care, ability to undertake usual activities, pain and discomfort, anxiety and depression), each with 5 levels of severity.
Sleep Quality - Pittsburgh Sleep Quality Index (PSQI) | Baseline (pre-intervention) and at follow-up 1(within in 48 hours of final treatment session, average of 3 weeks).
  The PSQI is a validated, self-reported questionnaire evaluating key areas including sleep duration, latency (how long it takes to fall asleep), efficiency, disturbances, use of sleep medication and day time dysfunction. Each section is scored individually, then added up to generate a global score ranging between 0-21. A score higher than 5 indicative of poor quality of sleep.
Usability - System Usability Scale (SUS) | Follow-up 1(within in 48 hours of final treatment session, average of 3 weeks).
  The SUS is a widely used 10 item questionnaire to measure how usable or user-friendly a system, product or service is.
Satisfaction - Quebec User Evaluation of Satisfaction with assistive Technology (QUEST) | Follow-up 1(within in 48 hours of final treatment session, average of 3 weeks).
  The QUEST questionnaire is a standardised 12-item, validated questionnaire designed to measure how satisfied users are with both their assistive devices and the service the received.
Cybersickness in VR Questionnaire (CSQ-VR). | Immediately after treatment visit 1, 2, 3 and at follow-up 1(within in 48 hours of final treatment session, average of 3 weeks).
  The CSQ-RV questionnaire will be used to assess symptoms commonly caused by VR exposure, such a nausea and dizziness.

CONTACTS AND LOCATIONS:
Overall Officials: Anju Jaggi, MSc, Study Director — Royal National Orthopaedic Hospital
Locations (1):
- Royal National Orthopaedic Hospital, Middlesex, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No